CLINICAL TRIAL: NCT02979977
Title: Single-Arm Phase II Trial of Dual Inhibition of EGFR With Afatinib and Cetuximab With Correlative Studies in the Treatment of Advanced Squamous Cell Cancers of the Head and Neck
Brief Title: Dual Inhibition of EGFR With Afatinib and Cetuximab in the Treatment of Advanced Squamous Cell Cancers of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Comprehensive Cancer Network (Network); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608018260
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Cancers of the Head and Neck
MeSH Terms: interventions — Cetuximab; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Experimental): Advanced squamous cell carcinoma of the head and neck region, having previously been treated on a platinum based regimen or with an immune checkpoint inhibitor. Subjects will receive Afatinib dose 30 mg per day and weekly/bi-weekly intravenous cetuximab.
  Interventions: Drug: cetuximab; Drug: afatinib

INTERVENTIONS:
Drug: cetuximab — 30-60 minutes after the recommended pre-medications, cetuximab will be administered intravenously at a dose of 400mg/m2 on cycle 1, day 1 of treatment (loading dose) and at a dose of 250mg/m2 every 7 days (+/- 1 day) thereafter. Alternatively, patients can be treated at a dose of 500mg/m2 every 14 days (+/- 2 days).
  Other Names: Erbitux
Drug: afatinib — Patients will take a single oral dose of afatinib each day at a dose of 30 mg. Afatinib dose will not be escalated beyond the 30 mg daily oral dose; dose reductions of afatinib can occur to manage treatment related adverse events.
  Other Names: GIOTRIF or GILOTRIF

SUMMARY:
This is a single arm Phase II study for patients with recurrent or metastatic squamous cell carcinoma of the head and neck, who are previously treated with a platinum based regimen or with an immune checkpoint inhibitor. The primary objective is to evaluate the efficacy of the combination of cetuximab and afatinib.

DETAILED DESCRIPTION:
This study will be a multicenter, single-arm, open-label Phase II trial. Patients with advanced squamous cell carcinoma of the head and neck, who are previously treated with a platinum based regimen or with immune checkpoint inhibitor therapy or both, will be eligible for participation on the study. After a baseline evaluation and biopsy (where feasible), they will be treated with weekly/bi-weekly intravenous cetuximab and daily oral afatinib. Biopsy will be repeated where feasible after 4 weeks (window of +1 week) on therapy and again at disease progression or end of treatment.

Treatment will continue until disease progression or development of Grade 3 or higher drug related toxicities that fail to resolve to Grade 2 despite appropriate supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck that is metastatic, recurrent or locally advanced and not treatable with curative intent.
* Previous treatment with a platinum-based regimen or immune checkpoint inhibitor or both.2-week washout period prior to treatment start will be required.
* Patients who have experienced progression of disease within 6 months following completion of a platinum-based chemoradiation in the definitive or adjuvant setting will be permitted.
* Prior cetuximab permitted if it was given as part of multi-modality therapy for initial treatment of locally advanced disease.
* Measurable disease based on RECIST v 1.1. Baseline measurements and evaluations must be obtained within 4 weeks of enrollment. Disease in previously irradiated sites is considered measurable if there has been unequivocal disease progression or biopsy-proven residual carcinoma following radiation therapy.
* ECOG performance status ≤2
* Adequate organ function, defined as all of the following:
* Hemoglobin ≥ 8 g/dl.
* Absolute neutrophil count (ANC) ≥1000 / mm3.
* Platelet count ≥75,000 / mm3.
* Estimated creatinine clearance > 45ml / min.
* Total Bilirubin ≤ 1.5 times upper limit of (institutional/central) normal (Patients with Gilbert's syndrome total bilirubin must be ≤4 times institutional upper limit of normal).
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤ three times the upper limit of (institutional/central) normal (ULN) (if related to liver metastases ≤ five times ULN).
* Ability to understand and the willingness to sign a written informed consent that is consistent with ICH-GCP guidelines.
* Negative urine or serum pregnancy test for women of childbearing potential
* A second eligibility review will always be provided by a Head and Neck Research Team associated for the New Haven Campus and a third review will be provided by the PI.

Exclusion Criteria:

* Prior erlotinib, gefitinib or lapatinib therapy or prior exposure to any investigational EGFR or panErbB reversible or irreversible inhibitor or any prior panitumumab or investigational EGFR-directed monoclonal antibody. Cetuximab is permitted if used for locally advanced disease, as long as no disease progression within 6 months. Cetuximab use is not permitted for recurrent/metastatic disease
* Radiotherapy within 2 weeks prior to enrollment. Palliative radiation to target organs may be allowed up to 2 weeks prior to enrollment, as long as there are other target lesions that can be monitored for response to study treatment.
* Known hypersensitivity to afatinib or its excipients
* Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control prior to study entry, for the duration of study participation and for at least 4 weeks after treatment has ended.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug.
* Concomitant malignancies at other sites that are being actively treated with systemic therapy
* Requiring treatment with any of the prohibited concomitant medications that cannot be stopped for the duration of trial participation.
* Clinically significant interstitial lung disease.
* Known history of untreated viral hepatitis or HIV.
* Patients with parenchymal brain metastases are not eligible, unless they have completed local therapy
* Leptomeningeal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2026-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Bhatia, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 50
Off Treatment | 49
Completed | 41
Not Completed | 9
Not completed — Death | 5
Not completed — Disease Progression | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 50 consented participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 63 [59 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 43
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 50
P16 Status [Count of Participants; unit: Participants]
  Negative | 29
  Positive | 21
Prior Lines of Treatment [Count of Participants; unit: Participants]
  Platinum | 49
  Anti-PD-1 | 37

OUTCOME MEASURES:

1. Primary Outcome: Tumor Shrinkage
Description: Objective Response Rate (Complete Response + Partial Response), defined by tumor shrinkage (mm), per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. RECIST v1.1 Response Categories are as follows: Complete Response (CR) - all pathological lymph nodes must be < 10 mm in short axis; Partial Response (PR) - at least a 30% decrease in the sum of diameters of target lesions; Stable Disease (SD) - The cancer has neither clearly improved nor worsened. Progressive Disease (PD) - at least a 20% increase in the sum of diameters of target lesions AND an absolute increase of ≥ 5 mm.
Time Frame: Disease progression or end of treatment (up to 2 years)
Population: Those who were response-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 47
Participants
  Complete Responses (CR) | 2
  Partial Response (PR) | 9
  No Response | 36
Statistical Analysis 1: Comparison: All Subjects; Test type: Superiority; Regression, Cox; Odds Ratio (OR) = 23.4, 95% CI 2-sided [12.3 to 38.0]

2. Secondary Outcome: Progression-free Survival in Months
Description: We will use Kaplan-Meier survival analysis to estimate the median PFS in the cohort. Data are presented by P16 status. The outcome measure title was updated to present the data in months, as analyzed, instead of weeks as originally registered.
Time Frame: 1 year follow-up
Population: Those that were response evaluable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 47
months
  P16 Negative: number analyzed (Participants) | 26
  P16 Negative | 3.8 [2.1 to NA] — Not enough events to calculate the upper bound CI.
  P16 Positive: number analyzed (Participants) | 21
  P16 Positive | 7.5 [4.8 to 12]

3. Secondary Outcome: Overall Survival in Months
Description: Measured by a monthly phone calls. We will use Kaplan-Meier survival analysis to estimate the median and OS in the cohort.
Time Frame: 1 year follow-up
Population: Those with an evaluable response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 47
months | 7.5 [4.8 to 12.0]

4. Secondary Outcome: Duration of Response in Weeks
Description: Presented is the time from treatment onset until best response.
Time Frame: Up to 6 years
Population: Only in those with a measurable response.
Measure: Median (Full Range); unit: weeks
Arm/Group | All Subjects
Number analyzed (Participants) | 11
weeks | 20.4 [1.0 to 293.4]

5. Secondary Outcome: Toxicity Assessed With National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Presented are a count of those that experienced at least 1 adverse event. Adverse event details are presented in the Adverse Events module.
Time Frame: Up to 2.5 years
Population: All those consented.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Participants | 49

6. Other Pre Specified Outcome: Exploratory Biomarker Analysis
Description: Analysis of tumor-tissue from biopsies obtained at baseline, after four weeks of treatment with the combination, and again at disease progression or end of treatment
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2.5 years
Description: All cause mortality is reported as death within 2.5 years of participants being placed on study.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 44/50
Serious Adverse Events (participants affected / at risk) | 20/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=50)
Dysphagia (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 2
Oral hemorrhage (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Infusion related reaction (General disorders) | 2
Pain (General disorders) | 1
Larygeal Edema (General disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Skin infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cancer of new histology (Investigations) | 1
Skin peeling (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=50)
Anemia (Blood and lymphatic system disorders) | 18
Lymphocyte count decreased (Blood and lymphatic system disorders) | 9
Sinus tachycardia (Cardiac disorders) | 4
Diarrhea (Gastrointestinal disorders) | 24
Mucositis oral (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 15
Pain (General disorders) | 6
Infusion related reaction (General disorders) | 6
Paronychia (Infections and infestations) | 7
Skin infection (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 3
Weight loss (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 35
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 8
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT02979977/Prot_SAP_000.pdf